CLINICAL TRIAL: NCT00635882
Title: A 2-Week Double-Blind, Placebo-Controlled, Parallel Group Study Comparing the Anti-Inflammatory Effects of Low, Medium, and High Dose Mometasone Furoate/Formoterol Fumarate MDI Formulation and Medium Dose Mometasone Furoate DPI and MDI Formulations in Adults and Adolescents With Persistent Allergic Asthma
Brief Title: Asthma Study Comparing Anti-Inflammatory Effects of 3 Doses of Mometasone Furoate/Formoterol Fumarate and Medium Dose Mometasone Furoate (Study P05122 AM1)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05122
Record Dates: First submitted 2008-01-21; First posted 2008-03-14 (Estimated); Results first posted 2011-02-09 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2022-02

CONDITIONS: Asthma; Airway Inflammation
Keywords: mometasone; formoterol
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- MF/F MDI 100/10 mcg (Experimental)
  Interventions: Drug: mometasone furoate/formoterol 100/10 mcg
- MF/F MDI 200/10 mcg (Experimental)
  Interventions: Drug: mometasone furoate/formoterol 200/10 mcg
- MF/F MDI 400/10 mcg (Experimental)
  Interventions: Drug: mometasone furoate/formoterol 400/10 mcg
- MF DPI 200 mcg (Experimental)
  Interventions: Drug: MF DPI 200 mcg
- MF MDI 200 mcg (Experimental)
  Interventions: Drug: MF MDI 200 mcg
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mometasone furoate/formoterol 100/10 mcg — mometasone furoate/formoterol 100/10 mcg twice daily (BID) (two inhalations of MF/F 50/5 from a metered-dose inhaler) for 14 days
  Other Names: MF/F (SCH 418131)
  Arms: MF/F MDI 100/10 mcg
Drug: mometasone furoate/formoterol 200/10 mcg — mometasone furoate/formoterol 200/10 mcg twice daily (BID) (two inhalations of MF/F 100/5 from a metered-dose inhaler) for 14 days
  Other Names: MF/F 200/10 (SCH 418131)
  Arms: MF/F MDI 200/10 mcg
Drug: mometasone furoate/formoterol 400/10 mcg — mometasone furoate/formoterol 400/10 mcg twice daily (BID) (two inhalations of MF/F 200/5 mcg from a metered-dose inhaler) for 14 days
  Other Names: MF/F 400/10 (SCH 418131)
  Arms: MF/F MDI 400/10 mcg
Drug: MF DPI 200 mcg — MF DPI 200 mcg twice daily (BID) (one inhalation of MF DPI 200 mcg) for 14 days
  Other Names: mometasone furoate (SCH 32088)
  Arms: MF DPI 200 mcg
Drug: MF MDI 200 mcg — MF MDI 200 mcg twice daily (BID) (two inhalations of MF MDI 100 mcg) for 14 days
  Other Names: mometasone furoate (SCH 32088)
  Arms: MF MDI 200 mcg
Drug: Placebo — MF/F MDI placebo twice daily (BID) (2 inhalations)
  Arms: Placebo

SUMMARY:
This is a 2-week double-blind, placebo-controlled, parallel group study comparing the anti-inflammatory effects of low, medium, and high dose mometasone furoate/formoterol fumarate (MF/F) metered dose inhaler (MDI) formulation and medium dose mometasone furoate (MF) dry powder inhaler (DPI) and MDI formulations in adults and adolescents with persistent allergic asthma.

DETAILED DESCRIPTION:
This is a 2-week double-blind, placebo-controlled, parallel group study comparing the anti-inflammatory effects of low, medium, and high dose mometasone furoate/formoterol fumarate MDI formulation and medium dose mometasone furoate (MF) DPI and MDI formulations in adults and adolescents with persistent allergic asthma. An open-label run in period is to be followed by a double-blind treatment period.

A total of 90 subjects (15 per treatment) will be enrolled to ensure 12 subjects per treatment at the Day 14 evaluation, accounting for a 20% drop-out rate. A sample size of 12 subjects per treatment is required to detect a treatment difference of 28% in percent change of eNO at Day 14, assuming a pooled standard deviation of 20% with a power of 90%. These estimates are based on examination of eNO levels in asthmatic vs healthy subjects in an article written by S.A. Kharitonov et. al, 2003.

Subjects will be randomized to one of six treatment groups (MF/F MDI 100/10 mcg BID, MF/F MDI 200/10 mcg BID, MF/F MDI 400/10 mcg BID, MF DPI 200 mcg BID, MF MDI 200 mcg BID, or Placebo MDI BID) according to an Schering-Plough Research Institute (SPRI) computer-generated randomization schedule. Randomization will be performed in appropriately sized blocks using random numbers generated by statistical analysis software (SAS).

ELIGIBILITY:
Inclusion Criteria:

* To document asthma diagnosis, historical reversibility defined as an increase in absolute forced expiratory volume (in liters) in 1 second (FEV1) of >= 12% and >= 200 mL must have been performed within 12 months of Screening. For subjects without historical reversibility, one of the following methods can be used at the Screening Visit or at any time before the Baseline Visit:

  * Demonstration of an increase in absolute FEV1 of at least 12% and a volume increase of at least 200 mL within 15-20 minutes after administration of 4 inhalations of albuterol/salbutamol (total dose 360 to 400 mcg) or of nebulized short-acting beta agonist (SABA) (2.5 mg), if confirmed as standard office practice, OR
  * Demonstration of a peak expiratory flow (PEF) variability of more than 20% expressed as a percentage of the mean highest and lowest morning prebronchodilator PEF over at least 1 week, OR
  * Demonstration of a diurnal variation PEF of more than 20% based on the difference between the prebronchodilator (before taking albuterol/salbutamol) morning value and the postbronchodilator value (after taking albuterol/salbutamol) from the evening before, expressed as a percentage of the mean daily PEF value on any day during the open-label Run-in Period. {The calculation formula: Diurnal PEF Variation = Absolute [(highest of 3 readings, PM Post-bronchodilator (BD) PEF from prior evening) - (highest of 3 readings, AM Pre-BD from morning value)]/[(highest PM Post-BD + highest AM Pre-BD)/2] * 100}
* At Screening and Baseline Visits, a subject must have persistent allergic asthma with an FEV1 >65% predicted.
* A subject must be allergic to at least one common allergen (grasses, trees, weeds, house dust mites, molds, dog and cat) as demonstrated by clinical symptoms when exposed to the allergen(s), and by skin prick testing or a radioallergosorbent (RAST) class >1 (excluding modified RAST procedure [mRAST]) within 2 years of inclusion in the study.
* If, based upon the medical judgment of the investigator, there is no inherent harm in changing the subject's current asthma therapy, the subject and/or parent/guardian) must agree to discontinue prescribed inhaled corticosteroid (ICS), anticholinergics, leukotriene receptor inhibitors, and long-acting beta-2 agonists at the Screening Visit as per required washouts, and be transferred to treatment with SABA for relief for 2 weeks before the Baseline/Randomization Visit.
* Clinical laboratory tests (complete blood count, blood chemistries, and urinalysis) conducted at the Screening Visit must be within normal limits or clinically acceptable to the investigator.
* An electrocardiogram (ECG) performed at the Screening Visit or within 30 days prior to Screening Visit must be clinically acceptable to the investigator and have a QTc interval <440 milliseconds for males and <450 msec for females.
* At Screening or any time prior to Baseline, a subject must have an eNO level of >30 parts per billion (ppb) at a flow rate of 50 mL/second.
* At Screening or any time before Baseline, a subject must have a sputum eosinophil count >3% of total cell count.
* Willingness to give written informed consent and ability to adhere to dose and visit schedules. A subject 12 to 17 years of age must also provide written assent.
* A nonpregnant female subject of childbearing potential (with a negative serum pregnancy test at Screening) must use a medically acceptable, adequate form of birth control. If not currently sexually active she must agree to use a double-barrier method if she becomes sexually active during the study.

Exclusion Criteria:

* Use of systemic glucocorticosteroids within 3 months before Screening.
* Upper or lower respiratory tract infection within 4 weeks before Screening.
* Decrease in absolute FEV1 >20% between Screening and Baseline Visits.
* Requirement for > 8 inhalations per day of SABA MDI, or 2 or more nebulized treatments of 2.5 mg SABA, on any 2 consecutive days between the Screening and Baseline Visits.
* A decrease in AM or PM PEF below the Run-in Period stability limit on any 2 consecutive days before Baseline. At Visit 1, the Run-in Period stability limit for PEF will be established based on the subject's personal best. If the subject does not have a historical personal best, the historical PEF measurement will be the PEF predicted based on the subject's sex, age, and height. PEF value to be multiplied by 0.70 to determine stability limit.
* A clinical asthma exacerbation defined as a clinical deterioration of asthma that results in emergency treatment, hospitalization for asthma, or treatment with additional, excluded asthma medication (including oral or other systemic corticosteroids but allowing SABA), as per investigator, between Screening and Baseline Visits.
* Inability to induce sputum after 1 or 2 trys.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nolte H, Pavord I, Backer V, Spector S, Shekar T, Gates D, Nair P, Hargreave F. Dose-dependent anti-inflammatory effect of inhaled mometasone furoate/formoterol in subjects with asthma. Respir Med. 2013 May;107(5):656-64. doi: 10.1016/j.rmed.2013.02.010. Epub 2013 Mar 13. PMID 23490226

RESULTS

PARTICIPANT FLOW:
Groups:
- MF/F MDI 100/10 mcg: Mometasone furoate/formoterol fumarate (MF/F) metered dose inhaler (MDI) 100/10 mcg twice daily (BID) for 14 days
- MF/F MDI 200/10 mcg: MF/F MDI 200/10 mcg BID for 14 days
- MF/F MDI 400/10 mcg: MF/F MDI 400/10 mcg BID for 14 days
- MF DPI 200 mcg: Mometasone furoate (MF) dry powder inhaler (DPI) 200 mcg BID for 14 days
- MF MDI 200 mcg: MF MDI 200 mcg BID for 14 days
- Placebo: Placebo MDI BID for 14 days
Period: Overall Study
Arm/Group | MF/F MDI 100/10 mcg | MF/F MDI 200/10 mcg | MF/F MDI 400/10 mcg | MF DPI 200 mcg | MF MDI 200 mcg | Placebo
Started | 20 | 17 | 12 | 15 | 16 | 13
Completed | 19 | 17 | 12 | 15 | 16 | 13
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MF/F MDI 100/10 mcg | MF/F MDI 200/10 mcg | MF/F MDI 400/10 mcg | MF DPI 200 mcg | MF MDI 200 mcg | Placebo | Total
Number analyzed (Participants) | 20 | 17 | 12 | 15 | 16 | 13 | 93
Age, Customized [Number; unit: participants]
  18 to <65 years | 20 | 14 | 11 | 15 | 16 | 11 | 87
  > or = to 65 years | 0 | 3 | 1 | 0 | 0 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 4 | 6 | 6 | 8 | 47
  Male | 7 | 7 | 8 | 9 | 10 | 5 | 46

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline to Day 14 in Exhaled Nitric Oxide (eNO) Parts Per Billion (Ppb)
Time Frame: Baseline to Day 14
Population: All Randomized Participants
Measure: Mean (Standard Deviation); unit: percentage of eNO
Arm/Group | MF/F MDI 100/10 mcg | MF/F MDI 200/10 mcg | MF/F MDI 400/10 mcg | MF DPI 200 mcg | MF MDI 200 mcg | Placebo
Number analyzed (Participants) | 19 | 16 | 12 | 14 | 15 | 13
percentage of eNO | -35.3 (40.3) | -45.4 (40.3) | -61.4 (40.3) | -51.3 (40.3) | -46.1 (40.3) | 0.1 (40.3)
Statistical Analysis 1: Comparison: MF/F MDI 400/10 mcg vs Placebo; Analysis of covariance (ANCOVA) model with treatment and baseline eNO as a covariate was used. Standard deviation is a Pooled Standard deviation from ANCOVA Model with treatment effect and baseline eNO as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg vs Placebo; ANCOVA model with treatment and baseline eNO as a covariate was used. Standard deviation is a Pooled Standard deviation from ANCOVA Model with treatment effect and baseline eNO as a covariate; Test type: Superiority or Other; p = 0.003, ANCOVA
Statistical Analysis 3: Comparison: MF/F MDI 100/10 mcg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.018, ANCOVA

2. Secondary Outcome: Mean Percent Change From Baseline to Day 7 in eNO Ppb
Time Frame: Baseline to Day 7
Population: All Randomized Participants
Measure: Mean (Standard Deviation); unit: percentage of eNO
Arm/Group | MF/F MDI 100/10 mcg | MF/F MDI 200/10 mcg | MF/F MDI 400/10 mcg | MF DPI 200 mcg | MF MDI 200 mcg | Placebo
Number analyzed (Participants) | 19 | 16 | 12 | 14 | 15 | 13
percentage of eNO | -37.9 (36.3) | -39.7 (36.3) | -45.6 (36.3) | -46.0 (36.3) | -37.2 (36.3) | 4.8 (36.3)
Statistical Analysis 1: Comparison: MF/F MDI 400/10 mcg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.002, ANCOVA
Statistical Analysis 3: Comparison: MF/F MDI 100/10 mcg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.002, ANCOVA

3. Secondary Outcome: Mean Percent Change From Baseline to Day 14 in Sputum Eosinophil Count (Percentage)
Time Frame: Baseline to Day 14
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: percentage of Sputum Eosinophil Count
Arm/Group | MF/F MDI 100/10 mcg | MF/F MDI 200/10 mcg | MF/F MDI 400/10 mcg | MF DPI 200 mcg | MF MDI 200 mcg | Placebo
Number analyzed (Participants) | 15 | 13 | 7 | 12 | 11 | 10
percentage of Sputum Eosinophil Count | 21.1 (127.6) | -35.5 (127.6) | -75.4 (127.6) | -55.3 (127.6) | -33.7 (127.6) | 71.7 (127.6)
Statistical Analysis 1: Comparison: MF/F MDI 400/10 mcg vs Placebo; ANCOVA model with treatment and baseline eosinophils as a covariate was used. Standard deviation is a Pooled Standard deviation from ANCOVA Model with treatment effect and baseline EOS as a covariate; Test type: Superiority or Other; p = 0.024, ANCOVA
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.051, ANCOVA
Statistical Analysis 3: Comparison: MF/F MDI 100/10 mcg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.336, ANCOVA

4. Secondary Outcome: Mean Change From Baseline to Day 15 of Mannitol Challenge
Description: Mannitol challenge (also referred to as PD15) is the provocative dose of mannitol required to produce a 15% reduction in the forced expiratory volume (in liters) in one second (FEV1).
Time Frame: Baseline to Day 15
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | MF/F MDI 100/10 mcg | MF/F MDI 200/10 mcg | MF/F MDI 400/10 mcg | MF DPI 200 mcg | MF MDI 200 mcg | Placebo
Number analyzed (Participants) | 12 | 9 | 6 | 8 | 9 | 9
milligrams
  Baseline | 102.2 (106.7) | 48.6 (106.7) | 67.9 (106.7) | 137.6 (106.7) | 126.0 (106.7) | 159.4 (106.7)
  Mean Change from Baseline to Day 15 | 176.6 (264) | 153.8 (264) | 162.9 (264) | 159.4 (264) | 146.2 (264) | -63.7 (264)
Statistical Analysis 1: Comparison: MF/F MDI 400/10 mcg vs Placebo; ANCOVA model with treatment and baseline PD15 as a covariate was used. Standard deviation is a Pooled Standard deviation from ANCOVA Model with treatment effect and baseline PD15 as a covariate; Test type: Superiority or Other; p = 0.120, ANCOVA; Analysis applies to Mean Change from Baseline to Day 15
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.103, ANCOVA; Analysis applies to Mean Change from Baseline to Day 15
Statistical Analysis 3: Comparison: MF/F MDI 100/10 mcg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.048, ANCOVA; Analysis applies to Mean Change from Baseline to Day 15

5. Secondary Outcome: Change From Baseline in AM Total Asthma Symptom Score at Days 2-15
Description: Twice daily, participants rated the following asthma symptoms as experienced during the time period since the last evaluation: wheezing, difficulty breathing, and cough on a scale of 0 (none) to 3 (severe, very uncomfortable and interfered with most or all of normal daily activities/sleep). The total asthma symptom score ranged from 0 to 9. The results were recorded in the participant's diary.
Time Frame: Baseline and Days 2-15
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MF/F MDI 100/10 mcg | MF/F MDI 200/10 mcg | MF/F MDI 400/10 mcg | MF DPI 200 mcg | MF MDI 200 mcg | Placebo
Number analyzed (Participants) | 20 | 17 | 12 | 15 | 16 | 13
units on a scale
  Baseline | 1.6 (1.66) | 1.2 (1.66) | 2.2 (1.66) | 1.5 (1.66) | 1.1 (1.66) | 1.4 (1.66)
  Mean Change from Baseline to Days 2-15 | -0.7 (1.28) | -0.7 (1.28) | -1.5 (1.28) | -1.2 (1.28) | -0.5 (1.28) | -0.2 (1.28)
Statistical Analysis 1: Comparison: MF/F MDI 400/10 mcg vs Placebo; One-way analysis of variance (ANOVA) model with treatment effect was used. Standard deviation is a Pooled Standard deviation from the one-way ANOVA model with treatment effect; Test type: Superiority or Other; p = 0.018, ANOVA; Analysis applies to Mean Change from Baseline to Days 2-15
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg vs Placebo; One-way ANOVA model with treatment effect was used. Standard deviation is a Pooled Standard deviation from the one-way ANOVA model with treatment effect; Test type: Superiority or Other; p = 0.261, ANOVA; Analysis applies to Mean Change from Baseline to Days 2-15
Statistical Analysis 3: Comparison: MF/F MDI 100/10 mcg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.334, ANOVA; Analysis applies to Mean Change from Baseline to Days 2-15

6. Secondary Outcome: Change From Baseline in PM Total Asthma Symptom Score at Days 1-15
Description: as for outcome 5
Time Frame: Baseline and Days 1-15
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MF/F MDI 100/10 mcg | MF/F MDI 200/10 mcg | MF/F MDI 400/10 mcg | MF DPI 200 mcg | MF MDI 200 mcg | Placebo
Number analyzed (Participants) | 20 | 17 | 12 | 15 | 15 | 13
units on a scale
  Baseline | 1.7 (1.62) | 1.1 (1.62) | 2.1 (1.62) | 1.6 (1.62) | 1.6 (1.62) | 1.7 (1.62)
  Mean Change from Baseline to Days 1-15 | -0.4 (1.24) | -0.6 (1.24) | -1.4 (1.24) | -1.1 (1.24) | -0.7 (1.24) | -0.3 (1.24)
Statistical Analysis 1: Comparison: MF/F MDI 400/10 mcg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.037, ANOVA; Analysis applies to Mean Change from Baseline to Days 1-15
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.643, ANOVA; Analysis applies to Mean Change from Baseline to Days 1-15
Statistical Analysis 3: Comparison: MF/F MDI 100/10 mcg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.963, ANOVA; Analysis applies to Mean Change from Baseline to Days 1-15

7. Secondary Outcome: Change From Baseline in AM Peak Expiratory Flow (PEF) at Days 2-15
Time Frame: Baseline and Days 2-15
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | MF/F MDI 100/10 mcg | MF/F MDI 200/10 mcg | MF/F MDI 400/10 mcg | MF DPI 200 mcg | MF MDI 200 mcg | Placebo
Number analyzed (Participants) | 20 | 17 | 12 | 15 | 16 | 13
liters/minute
  Baseline | 452.6 (112.1) | 421.2 (112.1) | 468.7 (112.1) | 466.3 (112.1) | 473.3 (112.1) | 413.2 (112.1)
  Mean Change from Baseline to Days 2-15 | 48.1 (47.0) | 46.9 (47.0) | 69.8 (47.0) | 30.3 (47.0) | 30.8 (47.0) | -9.0 (47.0)
Statistical Analysis 1: Comparison: MF/F MDI 400/10 mcg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA; Analysis applies to Mean Change from Baseline to Days 2-15
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.002, ANOVA; Analysis applies to Mean Change from Baseline to Days 2-15
Statistical Analysis 3: Comparison: MF/F MDI 100/10 mcg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA; Analysis applies to Mean Change from Baseline to Days 2-15

8. Secondary Outcome: Change From Baseline in PM PEF at Days 1-15
Time Frame: Baseline and Days 1-15
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | MF/F MDI 100/10 mcg | MF/F MDI 200/10 mcg | MF/F MDI 400/10 mcg | MF DPI 200 mcg | MF MDI 200 mcg | Placebo
Number analyzed (Participants) | 20 | 17 | 12 | 15 | 15 | 13
liters/minute
  Baseline | 462.0 (114.6) | 437.2 (114.6) | 486.7 (114.6) | 484.4 (114.6) | 472.5 (114.6) | 422.7 (114.6)
  Mean Change from Baseline to Days 1-15 | 47.7 (42.3) | 34.5 (42.3) | 66.8 (42.3) | 20.2 (42.3) | 28.3 (42.3) | 4.5 (42.3)
Statistical Analysis 1: Comparison: MF/F MDI 400/10 mcg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA; Analysis applies to Mean Change from Baseline to Days 1-15
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.057, ANOVA; Analysis applies to Mean Change from Baseline to Days 1-15
Statistical Analysis 3: Comparison: MF/F MDI 100/10 mcg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.005, ANOVA; Analysis applies to Mean Change from Baseline to Days 1-15

9. Other Pre Specified Outcome: Baseline Exhaled Nitric Oxide (eNO) Parts Per Billion (Ppb)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | MF/F MDI 100/10 mcg | MF/F MDI 200/10 mcg | MF/F MDI 400/10 mcg | MF DPI 200 mcg | MF MDI 200 mcg | Placebo
Number analyzed (Participants) | 19 | 16 | 12 | 14 | 15 | 13
ppb | 54.8 (40.8) | 70.0 (40.8) | 77.1 (40.8) | 102.6 (40.8) | 66.2 (40.8) | 79.6 (40.8)

ADVERSE EVENTS:
Arm/Group | MF/F MDI 100/10 MCG BID | MF/F MDI 200/10 MCG BID | MF/F MDI 400/10 MCG BID | MF DPI 200 MCG BID | MF MDI 200 MCG BID | PLACEBO
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 0/12 | 0/15 | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 2/20 | 8/17 | 1/12 | 2/15 | 6/16 | 2/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF/F MDI 100/10 MCG BID (N=20) | MF/F MDI 200/10 MCG BID (N=17) | MF/F MDI 400/10 MCG BID (N=12) | MF DPI 200 MCG BID (N=15) | MF MDI 200 MCG BID (N=16) | PLACEBO (N=13)
EAR DISCOMFORT (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPINAL CORD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUNBURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish/present any interim results without prior

sponsor written consent. The investigator agrees to provide to the sponsor, 45 days prior to submission, review copies for publication that report any study results. The sponsor has the right to review and comment. If the parties disagree, investigator agrees to meet with the sponsor, prior to submission for publication, to discuss and resolve any such issues/disagreement.